CLINICAL TRIAL: NCT07281092
Title: Comparing Psychosocial Supports for Adolescents With ADHD: What Works Best for Whom and Why?
Brief Title: Comparative Efficacy of Organizational Skills Training (OST) and Mindfulness-Based Intervention (MBI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Margaret Sibley, Professor of Psychiatry & Behavioral Sciences, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005325
Record Dates: First submitted 2025-09-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: ADHD; ADHD - Attention Deficit Disorder With Hyperactivity
Keywords: adhd; attention deficit hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — TOPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organizational Skills Training (OST) (Experimental): Adolescents with an ADHD diagnosis (confirmed via SCH's electronic health record or an external documentation of a diagnosis) seeking treatment at the the Seattle Children's BAM clinic will be recruited. They will be randomized 1:1 to OST or MBI, which are both treatments that are offered as standard clinical care, billable treatments at the SCH BAM clinic. Adolescents and their caregivers will complete rating scales at pre-treatment and post-treatment remotely via Research Electronic Data Capture.
  Both treatments are eight 90 minute sessions and are offered as billable services by the SCH BAM clinic as a standard of care.
  Interventions: Behavioral: Organizational Skills Training
- Mindfulness-Based Intervention (MBI) (Experimental): Adolescents with an ADHD diagnosis (confirmed via SCH's electronic health record or an external documentation of a diagnosis) seeking treatment at the the Seattle Children's BAM clinic will be recruited. They will be randomized 1:1 to OST or MBI, which are both treatments that are offered as standard clinical care, billable treatments at the SCH BAM clinic. Adolescents and their caregivers will complete rating scales at pre-treatment and post-treatment remotely via Research Electronic Data Capture.
  Both treatments are eight 90 minute sessions and are offered as billable services by the SCH BAM clinic as a standard of care.
  Interventions: Behavioral: Mindfulness-Based Intervention

INTERVENTIONS:
Behavioral: Organizational Skills Training — OST is a treatment offered as standard clinical care, billable treatments at the SCH BAM Clinic. There are eight 90 minute long sessions.
  Other Names: TOPS
  Arms: Organizational Skills Training (OST)
Behavioral: Mindfulness-Based Intervention — MBI is a treatment offered as standard clinical care, billable treatments at the SCH BAM clinic. There are eight 90 minute long sessions
  Other Names: MAPA; MBI
  Arms: Mindfulness-Based Intervention (MBI)

SUMMARY:
This randomized control trial comparing Organizational Skills Training (OST) and Mindfulness-Based Intervention (MBI) among adolescents with a pre-existing ADHD diagnosis presenting to the Duke ADHD Program.

Both treatments are eight 90 minute sessions.

The research component will involve a pre-treatment assessment and post-treatment assessment. Both assessments will involve adolescents and one caregiver to complete questionnaires over REDCap. Rating scales will include ADHD symptom severity (Conners 3: self and parent report), functional impairment (IRS: self and parent report), executive functioning (BRIEF-2: parent report), emotion dysregulation (DERS: self and parent report), trait mindfulness (FFMQ: self report), organizational skills (BRIEF-2: parent report), treatment satisfaction (self report and parent report) and credibility (self report and parent report). Post-treatment assessments for feasibility will include attendance (measured over the course of treatment) and homework completion rates on a scale of 1 to 5 in which 5 indicates higher homework completion. We will also assess acceptability via individual items on a Likert scale (self report): overall satisfaction, how much was learned about ADHD, usefulness of information learned, content relevance to individual experience, comprehension of strategies, confidence about using strategies, likelihood of using strategies, helpfulness to share with the group, benefits from hearing from other group members, willingness to recommend the same treatment to others, and whether or not treatment was beneficial.

DETAILED DESCRIPTION:
This will be a randomized controlled trial in which incoming patients (N=36) who have been referred for ADHD psychosocial treatment at the Seattle Children's Behavior, Attention, Management clinic between ages 13-17 will be offered the opportunity to participate in this study.

If they wish to participate, they will be randomly assigned to receive the MAPA MBI or to receive Organization Skills Training (TOPS) at the clinic. Both groups will be 8-week, 90 groups that will run simultaneously via telehealth delivered by routine clinicians in the BAM clinic. Both groups will have one "pre-session" that parents join that explains the purpose of the group and what parents and teens can do to work together and support home practice of skills learned during the group. We will collect baseline and post-treatment ratings of outcome measures. There will be two cohorts (fall and winter and each cohort will enroll 18 youth for random assignment at a 1:1 ratio). Incoming patients who do not wish to participate in the study will still be eligible to enroll in standard psychosocial treatment groups at the BAM clinic that they would otherwise be eligible for (i.e., declining to participate will not delay the treatment they otherwise would receive in the clinic).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between the ages of 13-17 years
* Pre-existing diagnosis of ADHD in medical record
* Seeking treatment at the Seattle Children's Hospital BAM Clinic

Exclusion Criteria:

* Psychiatric comorbidity that interferes with treating ADHD as the presenting concern per the study team.
* Other concerns besides ADHD that would interfere with study participation according to the study team.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ADHD symptoms | From enrollment to the end of treatment at 8 weeks
  Measured using the Conners 3 self and parent reports from the pre- and post- treatment questionnaires. Participants will rate several statements using a scale ranging from 0 to 3 (from Not True at All to Very Much True). Higher scores indicate more behavioral, emotional, or ADHD-related concerns.
Functional Impairment | From enrollment to the end of treatment at 8 weeks.
  Measured using the Impairment Rating Scale [IRS]: self and parent reports from the pre-and post-treatment questionnaires. Each item rated 0-6; total or mean scores vary by scoring method, with higher scores indicating greater functional impairment.
Executive Functioning | From enrollment to the end of treatment at 8 weeks.
  Measured using Behavior Rating Inventory of Executive Functioning [BRIEF-2]: parent report from pre-and post-treatment questionnaires. Participants will rate several behaviors on a scale of 1-3 depending how often that behavior occurs. Higher scores indicate higher executive functioning difficulties.
Emotion Dysregulation | From enrollment to the end of treatment at 8 weeks.
  Measured using Difficulties in Emotion Regulation Scale [DERS]: self and parent reports from pre-and post-treatment questionnaires. Each item on the DERS is rated using a 5-point Likert scale, with higher scores indicating greater difficulties with emotional regulation.
Trait Mindfulness | From enrollment to the end of treatment at 8 weeks.
  Measured using the Five Facet Mindfulness Questionnaire [FFMQ]: self report given during the pre-and post-treatment questionnaires. Each item on the FFMQ is rated using a 5-point Likert scale, with a higher total score indicating greater mindfulness.
Organizational Skills | From enrollment to the end of treatment at 8 weeks.
  Measured using the Behavior Rating Inventory of Executive Functioning (BRIEF-2): parent report given during the pre- and post- treatment questionnaires. Participants will rate several behaviors on a scale of 1-3 depending how often that behavior occurs. Higher scores indicate higher executive functioning difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT07281092/Prot_SAP_000.pdf